CLINICAL TRIAL: NCT03165500
Title: Comparative Evaluation of Three Anxiety Control Protocols in Third Molar Extraction With Midazolam, Diazepam and Nitrous Oxide - Randomized Clinical Trial.
Brief Title: Comparative Evaluation of Three Anxiety Control Protocols in Third Molar Extraction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Michelle Bianchi de Moraes, Professor Assistente Doutor - Departamento de Diagnóstico e Cirurgia - São Paulo State University (Unesp), Institute of Science and Technology, São José dos Campos, Brasil., Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Universidade Estadual Paulista
Record Dates: First submitted 2017-05-17; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Anxiety Disease
Keywords: Exodontia; Sedation; Nitrous Oxide; Benzodiazepines
MeSH Terms: interventions — Diazepam; Midazolam; Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: The investigadors selected 120 third molars , with the need for exodontia, in patients aged 18 to 30 years, ASA I, and with moderate to high anxiety level according to the Corah Dental Anxiety Scale (DAS). Patients were randomly assigned to three groups of 40 patients and submitted to the following anxiety control protocol:
  * Group I - Sedation with 5 mg oral Diazepam 30 minutes before surgery;
  * Group II - Sedation with 7.5 mg oral Midazolam 30 minutes before surgery;
  * Group III - Inhaled sedation with a mixture of 40% of nitrous oxide and 60% of oxygen (Using the Porter MXR 3000 Flowmeter (Parker Hannifin - Hatfield, PA, Philadelphia)) started 5 minutes before surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diazepam (Active Comparator): Sedation of the anxious patient with diazepam 5 mg for measuring vital signs (blood pressure, heart rate, oxygen saturation) in the pre, trans and postoperative periods of third molar extraction.
  Interventions: Drug: Midazolam; Drug: Nitrous Oxide + Oxygen Gas; Procedure: Third molar extraction
- Midazolam (Active Comparator): Sedation of the anxious patient with midazolam 7.5 mg for measurement of vital signs (blood pressure, heart rate, oxygen saturation) in the pre, trans and postoperative periods of third molar extraction.
  Interventions: Drug: Diazepam; Drug: Nitrous Oxide + Oxygen Gas; Procedure: Third molar extraction
- Nitrous Oxide + Oxygen Gas (Active Comparator): Inhaled sedation of the mixture of 40% of nitrous oxide and 60% of oxygen gas for measurement of vital signs (blood pressure, heart rate, oxygen saturation) in the pre, trans and postoperative periods of third molar extraction.
  Interventions: Drug: Diazepam; Drug: Midazolam; Procedure: Third molar extraction

INTERVENTIONS:
Drug: Diazepam — Patients' vital signs (blood pressure, heart rate and oxygen saturation) were measured and recorded after 30 minutes of oral sedation with diazepam 5mg, during the extraction procedure and 15 minutes after the extraction.
  After the surgical procedure of extraction, the patients remained in recovery in the same room, being the criteria of discharge realized, from the normality of the vital signs and the response to the verbal commands, with the patient responsive and lucid.
  Other Names: Valium; Diazepam 5mg
  Arms: Midazolam; Nitrous Oxide + Oxygen Gas
Drug: Midazolam — Patients' vital signs (blood pressure, heart rate, and oxygen saturation) were measured and recorded after 30 minutes of oral sedation with midazolam 7.5mg during the extraction procedure and 15 minutes after the extraction.
  After the surgical procedure of extraction, the patients remained in recovery in the same room, being the criteria of discharge realized, from the normality of the vital signs and the response to the verbal commands, with the patient responsive and lucid.
  Other Names: Dormonid; Midazolam Oral Tablet
  Arms: Diazepam; Nitrous Oxide + Oxygen Gas
Drug: Nitrous Oxide + Oxygen Gas — Patients' vital signs (blood pressure, heart rate, and oxygen saturation) were measured and recorded after 30 minutes of sedation Inhalation with the mixture of 40% of nitrou oxide and 60% of oxygen, during the exodontia procedure and 15 minutes later.
  After the surgical procedure of extraction, the patients remained in recovery in the same room, being the discharge criteria performed, from the normality of the vital signs and the response to the verbal commands, with the patient responsive and lucid, and after the accomplishment of the test developed by Trieger et al.,(1971).
  Other Names: Nitrous Oxide; Nitrous Oxide Inhalant Product
  Arms: Diazepam; Midazolam
Procedure: Third molar extraction — Anxious patients in need of third molar extraction
  Other Names: Third molar surgery

SUMMARY:
The surgery for the extraction of the third molars is a procedure in Dentistry that generates a large picture of anxiety in the patient. One of the ways to try to soften this picture, are the professionals to use sedation. Thus, the objective of this study was to evaluate three sedation protocols, and to compare them with vital signs values, in order to obtain the sedation method with greater patients stability.

DETAILED DESCRIPTION:
The surgery for the extraction of third molars is one of the procedures in Dentistry that generates a great picture of anxiety in the patients, due to the expectation of pain and discomfort in the postoperative period, but mainly in the trans-operative period. One of the ways to try to minimize this situation is to use sedation, which is a relatively safe procedure performed by trained professionals and with an accurate indication for anxious patients. There are several protocols in the literature, but few comparative studies. Thus, the objective of this study was to evaluate three sedation protocols. For this purpose, 120 patients who required surgical treatment for extraction of third molars, aged between 18 and 30 years, and whose anxiety was moderate to severe according to the Corah Anxiety Scale from the School of Dentistry of São José Dos Campos (UNESP). These patients were randomly divided into three Groups: Group I - oral sedation with diazempam 5 mg; Group II - oral sedation with midazolam 7.5 mg and Group III - inhalation sedation with 40% of nitrous oxide . Prior to sedation, anxiety was quantified through the Corah Anxiety Scale. Vital signs (blood pressure, heart rate and oxygen saturation) were measured before sedation, after sedation, in the trans-operative period and 15 minutes after the end of sedation. The results will be submitted to descriptive statistics and compared using the statistical analysis of variance (ANOVA) and Tukey test with significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA1), without surgical contra indications, requiring avulsion of the included third and / or semi-molar third molars,
* Between the ages of 18 and 30,
* Patients who agreed to voluntarily participate in the research, after knowing the risks and benefits, and signing the Informed Consent Form (TCLE).
* Patients who presented moderate to high anxiety level in the questionnaire proposed by Corah in 1969.

Exclusion Criteria:

* Patients with any systemic or local change that contra indicated the procedure,
* Use of anti-inflammatories in the last 15 days,
* Pericoronitis,
* Patients who did not accept the Informed Consent Form (TCLE)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Assessment of blood pressure change | Immediately the arrival of the patient and before receiving sedation - 30 minutes after the patient receives oral sedation or 5 minutes after inhaled sedation- During the exodontia - 15 minutes after the end of surgery
  Evaluated in anxious patients submitted to the exodontia of third molars, sedated with diazepam, midazolam and nitrous oxide.The investigator evaluated with auscultatory instrument.

SECONDARY OUTCOMES:
Assessment of heart rate change | Immediately the arrival of the patient and before receiving sedation - 30 minutes after the patient receives oral sedation or 5 minutes after inhaled sedation- During the exodontia - 15 minutes after the end of surgery
  Evaluated in anxious patients submitted to the exodontia of third molars, sedated with diazepam, midazolam and nitrous oxide.The investigator evaluated with oscillometric monitor.
Assessment of oxygen saturation change | Immediately the arrival of the patient and before receiving sedation - 30 minutes after the patient receives oral sedation or 5 minutes after inhaled sedation- During the exodontia - 15 minutes after the end of surgery
  Evaluated in anxious patients submitted to the exodontia of third molars, sedated with diazepam, midazolam and nitrous oxide. The investigator evaluated with pulse oximeter

OTHER OUTCOMES:
Retrograde amnesia | Immediately the arrival of the patient and before receiving sedation - 30 minutes after the patient receives oral sedation or 5 minutes after inhaled sedation- 15 minutes after the end of surgery
  Evaluated in anxious patients submitted to the exodontia of third molars, sedated with diazepam, midazolam and nitrous oxide.Retrograde amnesia was evaluated by the investigator through the adapted test of Bulach et al., (2005), where 6 images were shown to the patient for a period of 5 seconds each
Test of Trieger | Measured 15 minutes after the end of surgery.]
  Evaluated in anxious patients submitted to the exodontia of third molars, sedated with nitrous oxide. Only for the patients in the group undergoing nitrous oxide sedation, the test developed by Trieger et al., (1971) was performed according to Malamed (2012). The researcher provides a drawing to the patient for the union of the points closest to the ideal.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle B Moraes, PHD, Principal Investigator — ICT-UNESP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joshi S, Ansari AS, Mazumdar S, Ansari S. A comparative study to assess the effect of oral alprazolam as premedication on vital parameters of patients during surgical removal of impacted mandibular third molars. Contemp Clin Dent. 2016 Oct-Dec;7(4):464-468. doi: 10.4103/0976-237X.194125. PMID 27994412
- [Result] Corah NL, Gale EN, Illig SJ. Assessment of a dental anxiety scale. J Am Dent Assoc. 1978 Nov;97(5):816-9. doi: 10.14219/jada.archive.1978.0394. PMID 31377
- [Result] Khader R, Oreadi D, Finkelman M, Jarmoc M, Chaudhary S, Schumann R, Rosenberg M. A prospective randomized controlled trial of two different sedation sequences for third molar removal in adults. J Oral Maxillofac Surg. 2015 Feb;73(2):224-31. doi: 10.1016/j.joms.2014.08.033. Epub 2014 Sep 16. PMID 25488309